CLINICAL TRIAL: NCT04572737
Title: Personalised Activity Plan for BREAKing UP Sitting Time in Patients With Peripheral Arterial Disease and Intermittent Claudication (The BREAK UP Study)
Acronym: BREAK UP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0795
Record Dates: First submitted 2020-09-14; First posted 2020-10-01 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Peripheral Arterial Disease
Keywords: intermittent claudication; exercise; physical activity; prolonged sitting; sedentary time
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: before and after intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Participants will take part in an 8-week home-based activity plan to break up sitting time by 60 minutes per day.
  Interventions: Behavioral: Activity plan to break up sitting time

INTERVENTIONS:
Behavioral: Activity plan to break up sitting time — This research study aims to prove efficacy of a home-based physical activity intervention targeted at reducing periods of prolonged sitting and improving physical function in patients with intermittent claudication.

SUMMARY:
Intermittent claudication is the most common manifestation of peripheral arterial disease, a common cardiovascular disease that causes blocked blood vessels (arteries) in the leg. Symptoms consist of persistent pain in one or both legs during exercise that is relieved with rest. Evidence suggests that high levels of uninterrupted sitting and sedentary behaviour are associated with cardiovascular disease risk, mortality and all-cause mortality. One of the main goals for treating people with intermittent claudication, is increased participation in physical activity. Supervised Exercise Programmes are recommended however these are not well tolerated and compliance is low. Alternative exercise, including short bouts of physical activity to break up sedentary time, has been suggested to help improve physical function.

This study will investigate whether alternative exercise, in the form of breaking up prolonged sitting time, will improve physical function in patients with intermittent claudication.

Patients will be screened during their routine clinic appointment at Glenfield Hospital. All other study activity will take place at the patients home.

Activity monitors will be worn for up to 8 days at baseline and follow-up, measuring step count and time, inactivity, activity time and intensity, and sleep duration. Participants will also be expected to wear activity monitors for the duration of the 8-week intervention to measure steps. Participants will be in the study for up to 18 weeks in total.

DETAILED DESCRIPTION:
Due to COVID-19 restrictions, the BREAK UP study is being conducted as an 8-week home-based before and after intervention study with the aim to improve physical function measured via the WIQ; and to reduce sitting time by up to 60 minutes per day, seven days a week.

Participants will be required to make contact with members of the research team twice to complete assessments remotely, once to complete a coaching consultation, and once per week during the 8-week activity plan to discuss their performance. Organisation of these, and any contact associated with recruitment may require more frequent contact with the research team via telephone or email.

Contact 1 (Recruitment/ eligibility):

Expression of interest to participate will be sought by the treating clinician at Glenfield hospital (listed on the delegation log), who will offer the patient a Participant Information Sheet, contact details form to complete and a consent form. The patient may then be approached by a member of the research team to take their consent, having read the information sheet, or if the participant is happy to be, a member of the research team will contact them within two weeks via telephone and/or email the participant to discuss the study in more detail and determine if they wish to participate or not. After which, they will be asked to complete the consent form and post this back to the research team. Once the signed and dated consent forms have been received, the researcher can organise for the baseline data to be collected.

Contact 2 (Baseline assessments):

Within 2 weeks participants will be required to complete baseline assessments which includes information on their date of birth/age, sex, ethnicity, smoking status, alcohol consumption, medical history (co-morbidities) and a number of questionnaires to assess their quality of life, breathlessness, anxiety and depression, fatigue and physical function. These will be completed over the telephone with the researcher or the researcher will post the questionnaires to the participants which will need to be completed and returned by post. These assessments will take approximately 1 hour.

Participants will also be posted two activity monitors (monitor 1 and 2) one of which will be wrist worn and the other thigh worn, as well as information on how to fit these. Participants will wear these for a period of up to 8 days to collect habitual physical activity data. A daily sleep-wake log will be used to collect data on participants sleep and wake-time, which will be posted, along with instructions on how to complete these, and returned via post along with the activity monitors.

Contact 3 (Coaching consultation):

Within 2 weeks participants will receive a telephone or video call which will be termed a "coaching consult", during which fourteen 2-minute activities to break sitting time will be discussed with a member of the research team. Video tutorials and/or instruction cards of these activities will be sent via post prior to the coaching consult. These activities and data from the habitual physical activity measure will be used to inform personalised activity plans whereby participants will be encouraged, using Bandura's social cognitive theory, to use these activities to reduce sitting time by up to 60 minutes per day for 8-weeks. This contact will take approximately 15 minutes. The 8-week activity plan will be prescribed, to complete at home and will begin within 2 weeks of this contact.

Participants will wear a wrist-worn activity monitor for the duration of the home-based 8-week intervention (monitor 3). They will be instructed on how to use these during the coaching consultation and how to complete daily diaries for monitor wear and activity completion for the 8-week period.

During the 8-week intervention participants will be contacted once a week via telephone or video to discuss their performance on the activity plan and completion of the daily diary. This will take approximately 15 minutes a week. A member of the research team will organise this over email or telephone.

A second 8-day habitual physical activity measurement period will take place during week 8 of the intervention. Activity monitors 1 and 2 will be posted to participants in good time along with instructions on how to fit these. During this second habitual physical activity measurement period participants will continue to wear wrist-worn activity monitor 3 as well.

Contact 4 (Follow-up):

Participants will then be contacted for their final assessments within one week of the end of the 8-week intervention. The follow-up assessments will include the same assessments as at baseline, except for one questionnaire, and will be completed via telephone with a member of the research team, or a researcher will be post these out to the participant for completion. The assessments will take approximately 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age ≥18 years
* ABPI <0.9 or >1.4 at rest OR >20% decrease post exercise. When ABPI is >0.9 but there is clinical suspicion of PAD, other non-invasive tests, which may include imaging, will be used to confirm diagnosis.
* History of intermittent claudication (exercise induced, aching/cramping, pain affecting the lower limbs or buttocks, which subsides with rest)
* Able and willing to give informed consent
* Able to speak, read, and write English
* Able to undertake light physical activity

Exclusion Criteria:

* Individuals with type 1, gestational, or monogenic diabetes mellitus
* On insulin therapy
* Hospital admission in preceding 3 months
* Current or planned pregnancy, or breast feeding
* Contra-indications to exercise
* Participation in CTIMP currently and/or in preceding 3 months
* Already participating in a structured SEP
* Serious illness with life-expectancy < 1 year
* Previous major amputation
* Recent cardiovascular event (within the last 12 months)
* Comorbidity that the research team considered to be a contraindication to involvement in the study
* Unable to communicate in English
* Recent diagnosis or treatment for cancer (within 12 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
To investigate overall changes in sitting time | 8 weeks
  Measured using accelerometers (comparison of time spent sitting at baseline vs. follow-up assessed via acceleration)
The walking impairment questionnaire | 8 weeks
  Total score for 16 questions measuring walking distance, speed and stair climbing from 0 (worst/inability) to 4 (best/without limitations)

SECONDARY OUTCOMES:
To investigate overall changes in time spent performing physical activity | 8 weeks
  Measured using accelerometers (comparison of time spent performing physical activity at baseline vs. follow up assessed via mean acceleration mg/day )
To investigate overall changes in time spent in light physical activity | 8 weeks
  Measured using accelerometers (comparison of time spent in light physical activity at baseline vs. follow up assessed via acceleration mins/day)
To investigate overall changes in time spent in moderate physical activity | 8 weeks
  Measured using accelerometers (comparison of time spent in moderate physical activity at baseline vs. follow up assessed via acceleration mins/day)
To investigate overall changes in time spent in vigorous physical activity | 8 weeks
  Measured using accelerometers (comparison of time spent in vigorous physical activity at baseline vs. follow up assessed via acceleration mins/day)
To investigate overall changes in time spent in prolonged sitting | 8 weeks
  Measured using accelerometers (comparison of time spent sitting at baseline vs. follow-up assessed via acceleration)
To investigate overall changes in time spent in sleep | 8 weeks
  Measured using accelerometers (comparison of time spent sleeping at baseline vs. follow-up assessed via acceleration)
To investigate whether personalised activity breaks in sitting time improve quality of life | 8 weeks
  Measured using the Vascular Quality of Life (VascuQoL) questionnaire
To investigate whether personalised activity breaks in sitting time improve quality of life | 8 weeks
  Measured using the Euro Quality of Life (EQ-5D-5L) questionnaire
To investigate whether personalised activity breaks in sitting time improve breathlessness | 8 weeks
  Measured using the modified medical research council (mMRC) dyspnoea scale
To investigate whether personalised activity breaks in sitting time improve fatigue | 8 weeks
  Measured using Chalder's Fatigue Scale
To investigate whether personalised activity breaks in sitting time improve anxiety and depression | 8 weeks
  Measured using the hospital anxiety and depression scale

CONTACTS AND LOCATIONS:
Locations (1):
- J Perks, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Once we have analysed the results, we will present our findings at scientific meetings and publish in medical research journals. All these results will be anonymous, and it would not be possible to identify participants.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Perks J, Mcbride P, Rayt H, Payne T, Edwardson C, Rowlands AV, Messeder SJ, Yates T, Sayers R. Efficacy of a personalised activity plan for BREAKing UP sitting time in patients with intermittent claudication (the BREAK UP study). Diabetes Res Clin Pract. 2023 Oct;204:110925. doi: 10.1016/j.diabres.2023.110925. Epub 2023 Sep 28. PMID 37774979